CLINICAL TRIAL: NCT06756763
Title: Quality of Life After Head and Neck Free Flap Reconstruction: a Prospective Time to Deterioration Analysis
Brief Title: Head and Neck Quality of Life
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201402788B0
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Cancer; Free Flap
Keywords: Quality of life; Longitudinal; Survival
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Head and Neck Reconstruction patients: Head and Neck Reconstruction patients undergoing free flap reconstruction

SUMMARY:
This study examines the quality of life for patients after head and neck free flap reconstruction, both pre-operative and at least 1 year post-operative. It aims to find out what influences quality of life, and whether these changes are stable over time. It will use a new method of analysis called "Time to Deterioration" which tells us when a patient notices a significant change in their quality of life, when subsequently does not get better.

DETAILED DESCRIPTION:
Methods

Prospectively collected quality of life (QoL) study using a longitudinal TTD approach in a large cohort of head and neck free flap reconstruction patients. Questionnaires completed pre-operatively and at outpatient clinic visits, with concomitant examination and complication status recorded. Quality of life data collected by a clinician not involved in the research.

Participants and Setting Participants recruited from Chang Gung Memorial Hospital, Linkou, Taiwan. Inclusion criteria included all patients undergoing free flap reconstruction of benign or malignant head and neck disease, who had completed both pre-operative and a minimum of one post-operative questionnaire, at least 1 year post-operatively. Exclusion criteria included patients that did not undergo free flap reconstruction, extra-oral disease eg scalp, no pre-operative questionnaire, post-operative questionnaire without at least 1 year follow up, and patients unable to consent.

Primary outcome University of Winconsin Quality of Life (UW-QoL) questionnaire (Taiwan mandarin version v4) is a 12-item scale with additional global questions, scored from 0 to 100, with separate Physical and Social component scores providing a composite overall score.

Quality of Life primary outcomes Separate analysis of component scores, rather than overall score, is suggested in UW-QoL scoring guidelines. This study examined Physical component score as the primary outcome.

Missing data Missing data in UW QoL questionairres were handled according to published scoring guidelines, with a minimum 4 components in both physical and social subscores.

Time to Deterioration (TTD) definitions TTD methodology was used to assess changes in QoL over time. TTD is defined as a drop of > 5 points in QoL scores without a subsequent increase > 5 points compared to the previous score. Comparison with previous score accounts for 'response shift' in patient perceptions, whereby patients get accustomed to a new normal by internal recalibration. QoL studies typically use a General Linear Mixed Model approach that does not quantify for this 'response shift'. Using this approach also better accounts for 'reversibility' in QoL . Previous score was used rather than previous best score. An MCID of 5 points has been proposed for TTD methodology which is in line with estimates of 5-10% in the the UW QoL scoring guidelines.

Health Related Quality of Life (HRQoL) Deterioration Free Survival HRQoL deterioration free survival includes death (all cause death) as an event and is akin to overall survival.

ELIGIBILITY:
Inclusion Criteria:

* free flap reconstruction
* benign or malignant head and neck disease

Exclusion Criteria:

* did not undergo free flap reconstruction
* extra-oral disease eg scalp
* patients unable to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Head and neck disease both benign and maligant
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
University of Wisconsin Quality of Life Questionnaire | Once at enrollment pre-operatively, and repeated at least 1 year post-operatively
  University of Winconsin Quality of Life (UW-QoL) questionnaire (Taiwan mandarin version v4) is a 12-item scale with additional global questions, scored from 0 to 100, with separate Physical and Social component scores providing a composite overall score. Higher scores indicate higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
IPD shared on reasonable request to the authors